CLINICAL TRIAL: NCT00576329
Title: Topical 0.4% Ketorolac for the Inhibition of Miosis During Vitreoretinal Surgery: a Randomized, Placebo-controlled, Double-masked Study
Brief Title: Topical 0.4% Ketorolac and Vitreoretinal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Stephen Kim, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00000517
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Surgery
Keywords: vitreoretinal surgery, ketorolac, Acular, mydriasis
MeSH Terms: conditions — Mydriasis | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Ketorolac
- B (Experimental)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Topical use before surgery
  Other Names: Acular LS

SUMMARY:
To determine whether use of topical 0.4% ketorolac has any effect on pupil size during vitreoretinal surgery.

DETAILED DESCRIPTION:
Other outcomes will be to assess postoperative pain and inflammation and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18, routine elective vitrectomy

Exclusion Criteria:

* history of trauma, uveitis, prior intraocular surgery within 3 months, requirement of mechanical pupil dilation, prior inclusion of other eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in pupil size during vitreoretinal surgery | Surgery

SECONDARY OUTCOMES:
Postoperative pain and inflammation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Emory University
Locations (1):
- Emory Eye Clinic, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kim SJ, Lo WR, Hubbard GB 3rd, Srivastava SK, Denny JP, Martin DF, Yan J, Bergstrom CS, Cribbs BE, Schwent BJ, Aaberg TM Sr. Topical ketorolac in vitreoretinal surgery: a prospective, randomized, placebo-controlled, double-masked trial. Arch Ophthalmol. 2008 Sep;126(9):1203-8. doi: 10.1001/archopht.126.9.1203. PMID 18779478